CLINICAL TRIAL: NCT00297128
Title: Preoperative Chemoradiation With Capecitabine and Cetuximab Within a Multidisciplinary Therapeutic Approach in Patients With Operable T3-T4 Rectal Cancer: a Phase II Study
Brief Title: Preoperative Chemoradiation With Capecitabine and Cetuximab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Austrian Breast & Colorectal Cancer Study Group (Network)
Collaborators: Hoffmann-La Roche (Industry); Merck Gesellschaft mbH, Austria (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABCSG R03 (96) / TAKO 06
Record Dates: First submitted 2006-02-27; First posted 2006-02-28 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Rectal Cancer
Keywords: pilot study; rectal; cancer; phase II; preoperative; chemoradiation; capecitabine; cetuximab; operable; T4; ABCSG; TAKO; R03; 96; 06
MeSH Terms: conditions — Rectal Neoplasms; Neoplasms | interventions — Capecitabine; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator)
  Interventions: Drug: Capecitabine; Drug: Cetuximab

INTERVENTIONS:
Drug: Capecitabine — 825 mg/m2 bid (on each therapy day of first 4 therapy weeks)
  Other Names: Xeloda
Drug: Cetuximab — 400mg/m2 week 1, 250mg/m2 week 2-4
  Other Names: Erbitux

SUMMARY:
* feasibility and tolerance of preoperative therapy with Cetuximab in combination with Capecitabine and radiotherapy for patients with locally advanced operable rectal carcinoma
* collection of response rate (T-downstaging, pathological complete remission), correlation of responsiveness with EGFR-status

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80
* bioptical confirmed adenocarcinoma of the rectum in operable T3-T4NxM0 status. In spite of infiltration of the neighbouring organs the tumor has to be basically surgically complete resectable
* no former chemotherapy, radiotherapy of pelvis or abdomen and/or tumor resection of a rectum carcinoma
* WHO performance status 0-2
* adequate bone marrow reserve (granulocytes - not more than 1.500/µl; thrombocytes - not more than 100.000/µl)
* adequate hepatic function ( bilirubin - not more than 1.5 x ULN; GOT and GPT - not more than 3.5 x ULN)
* adequate renal function (creatinin - not more than 1.5 mg/dl)
* women of childbearing potential: exclusion of pregnancy (negative urin or serum pregnancy test)
* willingness of women of childbearing potential and accordingly of potent men to use approved contraceptives (e.g. birth-control pill, loop, condom) during and at least 3 month after conclusion of the study
* life expectancy of at least 3 month
* signed Informed Consent before recruitment
* exclusion of distant metastases at the time of recruitment

Exclusion Criteria:

* former radiotherapy of pelvis or abdomen
* former chemotherapy
* any other kind of malign tumor (except adequate treated skin basalioma or in situ cervical carcinoma) in the last 5 years
* general contraindication or known hypersensitivity against Cetuximab and/or Capecitabine
* Non malign disease, if there is a contraindication with radiotherapy or chemotherapy with Cetuximab and Capecitabine or a resection of the rectum: high-graded cardiac insufficiency, angina pectoris, hypertension or arrhythmia, hepatic disease, significant neurological or psychiatric disorders
* florid, serious infections at the time of recruitment
* legally limited contractual capability or evidence of neurological or psychiatric disease, if it will constrict the patients compliance in the opinion of the investigator
* evidence of lacking cooperation of the patient
* pregnant or breast feeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-10; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
feasibility and tolerance of preoperative therapy with Cetuximab in combination with Capecitabine and radiotherapy for patients with locally advanced operable rectal carcinoma | descriptive evaluation

SECONDARY OUTCOMES:
collection of response rate (T-downstaging, pCR), correlation of responsiveness with EGFR-status | description evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Josef Thaler, MD, Principal Investigator — Austrian Breast & Colorectal Cancer Study Group; Joerg Tschmelitsch, MD, Principal Investigator — Austrian Breast & Colorectal Cancer Study Group; Alexander de Vries, MD, Principal Investigator — Austrian Breast & Colorectal Cancer Study Group
Locations (10):
- Austria (10):
  - Hospital BHB St. Veit/Glan, Surgery, Saint Veit A. D. Glan, Carinthia
  - Hospital Wiener Neustadt, Surgery, Wiener Neustadt, Lower Austria
  - Paracelsus Medical University Salzburg - Oncology, Salzburg, Salzburg
  - Medical University of Graz, Oncology, Graz, Styria
  - State Hospital Leoben, Leoben, Styria
  - Medical University of Innsbruck, Surgery, Innsbruck, Tyrol
  - Hospital BHS Linz, Radiooncology, Linz, Upper Austria
  - Klinikum Wels-Grieskirchen, Wels, Upper Austria
  - Medical University of Vienna, Radiotherapy, Vienna, Vienna
  - State Hospital Feldkirch, Feldkirch, Vorarlberg

REFERENCES:
- See also: Related Info — http://www.abcsg.at/